CLINICAL TRIAL: NCT00004387
Title: Phase II Double Blind Controlled Trial of Nigral Grafting in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Icahn School of Medicine at Mount Sinai (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/12102; MTS-94339; MTS-GCO-94-339
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Parkinson Disease; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Procedure: fetal nigral transplantation

SUMMARY:
OBJECTIVES:

I. Determine the effectiveness of fetal nigral transplantation in patients with Parkinson's disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a placebo controlled, randomized, double blind study. Patients are randomly assigned to 1 of 3 treatment groups. All patients receive 2 separate operations in which the substantia nigra from either 4 fetuses (Group A) or 1 fetus (Group C) is implanted into the striatum of each side.

Group B patients receive 2 separate placebo operations without fetal transplantation.

The second surgical procedure begins approximately 1 week after the first operation.

After 2 years, treatments are compared. If transplant is shown to benefit Parkinson's disease, then patients who received placebo operation will be offered transplant surgery in the final year of the study.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Advanced Parkinson's disease Hoehn-Yahr stage IV or worse during "off" periods Hoehn-Yahr stage III or better during "on" periods Predictable motor fluctuations with at least 20% of waking day in the "off" stage No atypical parkinsonism or secondary parkinsonism --Prior/Concurrent Therapy-- Biologic therapy: Not specified Chemotherapy: Stable doses of levodopa/carbidopa or any other antiparkinson therapy for 2 months prior to study Surgery: No previous intracranial/neurosurgical procedures --Patient Characteristics-- Renal: Creatinine clearance at least 70 mL/min or creatinine no greater than 1.8 mg/dL Protein no greater than 300 mg/dL Other: Not pregnant or nursing Adequate contraception required of fertile patients Prior history of good response to levodopa No sensitivity to cyclosporine Not HIV positive (e.g., HIV I or II) No human T-cell leukemia/lymphoma virus (HTLV-1) No tremors interfering with stereotactic surgery No clinically significant medical, neoplastic or infectious disease No clinically significant laboratory abnormality No dementia that precludes signing informed consent or score of less than 24 on Mini-Mental status examination

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 1996-01

CONTACTS AND LOCATIONS:
Overall Officials: C. Warren Olanow, Study Chair — Icahn School of Medicine at Mount Sinai